CLINICAL TRIAL: NCT01583894
Title: Multiple Areas of Pain (MAP): Epidemiology of Multisite Pain in the Chronic Pain Population
Brief Title: Multiple Areas of Pain (MAP)
Acronym: MAP
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A7003; CDM00044807 (Other: BSC protocol number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic pain patients

SUMMARY:
This study will collect pain-related information from chronic pain patients to gain an understanding of the prevalence of multi-site pain, and how it affects health outcomes like function, quality of life, depression, and anxiety.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic pain of the trunk and/or limbs lasting at least 6 months
* Overall pain intensity of at least 5 on a 0 to 10 scale
* Subject is able to independently complete all assessments in English
* 18 years of age or older
* Subject signs an Institutional Review Board-approved informed consent form provided in English

Key Exclusion Criteria:

* Currently implanted with an active implantable medical device to treat pain
* Currently exhibits any characteristic that renders the subject ineligible for current or future treatment with spinal cord stimulation for chronic pain of the trunk and/or limbs
* Subject has undergone an interventional pain procedure less than 1 month prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients resident in a US pain management practice.
Sampling Method: Non-Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Corporation
Locations (15):
- United States (15):
  - UCSD Medical Center - Jacobs Medical Center, La Jolla, California
  - Neurovations, Napa, California
  - Integrated Pain Specialists of Southern California, San Diego, California
  - Sheridan Clinical Research, Sunrise, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - Global Scientific Innovations - Advanced Pain Care Clinic, Evansville, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Comprehensive Pain & Rehabilitation, Pascagoula, Mississippi
  - Midwest Pain Center, Chesterfield, Missouri
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Channel Research, Pawleys Island, South Carolina
  - Houston Pain Associates, Houston, Texas
  - Nexus Pain Care, Provo, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Pain Patients: Patients suffering from chronic intractable pain of the trunk and/or limbs for a duration of at least 6 months
Period: Overall Study
Arm/Group | Chronic Pain Patients
Started | 828
Completed | 813
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: Patients suffering from chronic intractable pain of the trunk and/or limbs for a duration of at least 6 months
Arm/Group | Chronic Pain Patients
Number analyzed (Participants) | 828
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information available in 823 subjects
  years | 52.3 (13.23)
Sex/Gender, Customized [Number; unit: participants] — Gender information available in 826 subjects
  participants
    Female | 527
    Male | 299

OUTCOME MEASURES:

1. Primary Outcome: Multi-site Pain Index
Description: Multiple Site Pain Index (MSPI) was developed by collating multiple pain descriptors into a single index. Pain descriptors used for developing this index were percent body area in pain, number of painful areas, span of painful areas, and Regional Pain Ratings (RPRs) which includes data on pain severity and pain continuity for 47 body regions.
  MSPI score ranged from 0 to 1; 0 representing no pain and 1 representing extreme continuous pain over entire body, except the head and face regions.
Time Frame: single-visit
Population: MSPI was calculated using multiple pain descriptors which were obtained from pain drawings. 810 of the 813 patients that completed the study provided complete pain drawing data, and so MSPI could be calculated only in 810 patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain Patients
Number analyzed (Participants) | 810
units on a scale | 0.52 (0.13)

ADVERSE EVENTS:
Time Frame: Not applicable. Considering the non-interventional nature of this study, no adverse event data was collected.
Description: Considering the non-interventional nature of this study, no adverse event data was collected.
Arm/Group | Chronic Pain Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No